CLINICAL TRIAL: NCT03006835
Title: Different Dosage of Domestic and Imported Clopidogrel on the Platelet Inhibition Ratio in Patients Undergoing PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ky20162060-2
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Heart Disease
Keywords: Clopidogrel; Platelet Inhibition Ratio
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Investigator

ARMS (4):
- Domestic Clopidogrel 300mg (Experimental): Domestic Clopidogrel 300mg
  Interventions: Drug: Clopidogrel
- Domestic Clopidogrel 600mg (Experimental): Domestic Clopidogrel 600mg
  Interventions: Drug: Clopidogrel
- Imported Clopidogrel 300mg (Experimental): Imported Clopidogrel 300mg
  Interventions: Drug: Clopidogrel
- Imported Clopidogrel 600mg (Active Comparator): Imported Clopidogrel 600mg
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel

SUMMARY:
This is a single-center, randomized, single-blind, investigator-initiated, pharmacological study with a parallel design. Patients with non-ACS undergoing primary percutaneous coronary intervention will be randomized after informed consent, in a 1:1:1:1 ratio to the following treatment groups:

Group Α: Domestic Clopidogrel 300mg as a loading dose before PCI, followed by 75mg per day.

Group B: Domestic Clopidogrel 600mg as a loading dose before PCI, followed by 75mg per day.

Group B: Imported Clopidogrel 300mg as a loading dose before PCI, followed by 75mg per day.

Group D: Imported Clopidogrel 600mg as a loading dose before PCI, followed by 75mg per day.

Platelet inhibition ratio assessment by thrombelastogram will be performed，2 hours after the loading dose(Day 0)， 6 hours after thrombelastogram (Day 0), 30 day after thrombelastogram. Documentation of major adverse cardiac events (death, myocardial infarction, stroke, revascularization procedure with PCI or CABG) and serious adverse events (bleeding, other adverse events)will be performed until Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is scheduled to undergo non-urgent PCI
2. The patient is between 18 and 75 years of age (inclusive) and willing to comply with the protocol
3. The patient or legally acceptable representative is able to read and give written informed consent and has signed an informed consent form approved by the Investigator's IRB/IEC

Exclusion Criteria:

1. Estimated or measured weight < 55 kg
2. Acute non-ST-segment elevation myocardial infarction (NSTEMI) or ST-segment elevation myocardial infarction (STEMI) within 7 days prior to PCI
3. Uncontrolled hypertension at the time of initial study drug administration defined as measured systolic blood pressure > 190 mm Hg or diastolic blood pressure > 108 mm Hg
4. Patient has received a clopidogrel loading dose (≥300 mg) within 30 days prior to randomization; patients on maintenance clopidogrel may be enrolled
5. Administration of thrombolytic agents, fondaparinux, or oral anticoagulants (e.g., warfarin) within the 7 days prior to PCI
6. Estimated creatinine clearance (e.g. Cockcroft-Gault) < 45 mL/min
7. Anemia with hemoglobin level < 10 g/dL
8. Thrombocytopenia (platelet count < 100,000/mm3)
9. ALT and/or AST > 2.5 x the ULN or other indication of clinically significant hepatic dysfunction
10. Facial or head trauma within the last 30 days
11. Intraocular hemorrhage within the last 30 days
12. Gastrointestinal bleeding within the last 30 days
13. Active bleeding, or history of a bleeding disorder or known intracranial vascular malformation
14. Known allergy or contraindication to aspirin, heparin, clopidogrel, or to any contrast media
15. Participation in any investigational drug study within 30 days prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
ADP- induced platelet inhibition rate | 2 hours after the loading dose
ADP- induced platelet inhibition rate | 6 hours after the loading dose
ADP- induced platelet inhibition rate | 30 days after the loading dose

SECONDARY OUTCOMES:
R value (min) | 2 hours after the loading dose

CONTACTS AND LOCATIONS:
Overall Officials: ruining zhang, doctor, Study Director — Xijing Hospital, The Fourth Military Medical University, 15 Changle West Road, Xi'an, 710032, China